CLINICAL TRIAL: NCT05484128
Title: Lactobacillus Reuteri Strain Combination (Strains DSM 17938 and ATCC PTA 6475) in Children Treated With Proton Pump Inhibitors
Brief Title: Lactobacillus Reuteri Strain Combination in Children Treated With PPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Professor Ruggiero Francavilla, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROBPPI
Record Dates: First submitted 2021-11-25; First posted 2022-08-02 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Gastric Lesion; Proton Pump Inhibitor Adverse Reaction; Probiotic
Keywords: Reuteri; Proton Pump Inhibitor; gastrus; infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: randomized double bind with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: nobody knows the randomization code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastrus (Experimental): 86 patients Gastrus sachets/chewable caps: 2x108 CFU Lactobacillus reuteri DSM 17938 + 2x108 CFU Lactobacillus reuteri ATCC PTA 6475.
  Placebo sachets/chewable caps: Identical in shape, colour and taste to Gastrus capsules but without the Lactobacillus reuteri components.
  Both study products are delivered in identical containers. Dosing: Two sachets/cps twice a day. Length of treatment: Gastrus or placebo will be administered for all the duration of PPI administration (8 weeks) plus two weeks after its discontinuation. A final evaluation will be performed 4 weeks after the discontinuation of both Gastrus and placebo.
  Interventions: Dietary Supplement: Gastrus
- Placebo (Placebo Comparator): 86 patients Gastrus sachets/chewable caps: 2x108 CFU Lactobacillus reuteri DSM 17938 + 2x108 CFU Lactobacillus reuteri ATCC PTA 6475.
  Placebo sachets/chewable caps: Identical in shape, colour and taste to Gastrus capsules but without the Lactobacillus reuteri components.
  Both study products are delivered in identical containers. Dosing: Two sachets/cps twice a day. Length of treatment: Gastrus or placebo will be administered for all the duration of PPI administration (8 weeks) plus two weeks after its discontinuation. A final evaluation will be performed 4 weeks after the discontinuation of both Gastrus and placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Gastrus — Gastrus consisted of a mixture of two human strains of L. Reuteri DSM 17938 and ATCC PTA 6475.
  Gastrus will be administered for all the duration of PPI administration (8 weeks) plus two weeks after its discontinuation. A final evaluation will be performed 4 weeks after the discontinuation of both Gastrus.
  Arms: Gastrus
Other: Placebo — placebo has an identical preparation to Gastrus
  Arms: Placebo

SUMMARY:
Probiotics might be of help in preventing dysbiosis and emergence of SIBO. Gastrus consisted of a mixture of two human strains of L. Reuteri DSM 17938 and ATCC PTA 6475; the first have extensive data supporting its use in gastric infections (18) however, it lacks the anti-inflammatory properties that have been provided by L. Reuteri DSM ATCC PTA 6475 that has excellent acid resistance and has strong anti-inflammatory properties (19); for these reasons, Gastrus is the best candidate for this indication.

DETAILED DESCRIPTION:
Aim of study

Our aims are to assess if Gastrus administration:

1. reduces the incidence of SIBO;
2. reduces the risk of infections in children treated with gastric-acid inhibitors;
3. prevents perturbation of gut microbiota and related dysbiosis;

Study Product Gastrus sachets/chewable caps: 2x108 CFU Lactobacillus reuteri DSM 17938 + 2x108 CFU Lactobacillus reuteri ATCC PTA 6475.

Placebo sachets/chewable caps: Identical in shape, colour and taste to Gastrus capsules but without the Lactobacillus reuteri components.

Both study products are delivered in identical containers. Dosing: Two sachets/cps twice a day. Length of treatment: Gastrus or placebo will be administered for all the duration of PPI administration (8 weeks) plus two weeks after its discontinuation. A final evaluation will be performed 4 weeks after the discontinuation of both Gastrus and placebo.

Compliance, PP and ITT To be considered compliant the participant should have consumed at leas 80% of the doses. In order to improve compliance, the participants will be equipped with alarm-devices. Compliant patients will be assessed as Per-Protocol (PP). Patients that are non-compliant will be included in the Intention-To-Treat analysis.

Outcomes Primary efficacy parameter This study aimed at investigating if Gastrus administration prevents the emergence of SIBO and reduces the risk of infections in children treated with proton pump inhibitors and.

Exploratory parameters Ability of Gastrus to prevent and control gut microbiota alteration; Ability of Gastrus to improve GI symptoms for which the drug has been prescribed.

Sample size calculation Assuming that the average rate of infection in patient who assume PPI is 32% as compared to 9% of those who do not use the drug (16), to demonstrate an efficacy of the probiotic, keeping a power of the study of 80% and a p of 0,05 we need 78 patients for group that, considering a drop out of 10%, will became 86 per group (patient younger/older 4 years of age:0,75) This sample size is by far larger than needed to demonstrate the preventive effect on SIBO emergence.

ELIGIBILITY:
Inclusion Criteria:

* Age: children between 1 month and 14 years of age;

  o We start with children older than 4 years of age.
* Necessity of therapy with Proton Pump Inhibitors for Gastroesophageal reflux disease and/or Functional Dyspepsia;
* Informed consent obtained.

Exclusion Criteria:

* Neurological pathologies (PCI and Spastic tetra-paresis);
* Nasogastric feeding;
* Known immunodeficiency;
* Previous therapy with gastric acid inhibitors;
* HP infection;
* Assumption of prebiotics, other probiotics or symbiotics in the previous month;
* Malnutrition or severe dystrophy;
* Cystic Fibrosis.

Ages: 12 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Variation in Lactulose breath test results | at baseline and week 10
  This study aimed at investigating if Gastrus administration prevents the emergence of SIBO in children treated with proton pump inhibitors. This test will be performed to assess the presence of SIBO before PPI treatment and at week 10 (end of PPI treatment).
Variation in results of Health Questionnaire for Data Collection | at baseline and weekly until week 14
  A diary will be given to the parents, with instructions to report the following: systemic symptoms including fever, headache, restless, myalgia, irritability; gastrointestinal or respiratory symptoms; use of drugs (antibiotics, antipyretics, steroids); emergency department medical examinations; hospitalizations; possible adverse events; consumption of the study products; school days lost by the children; working days lost by the parents.

SECONDARY OUTCOMES:
fecal analysis | 14 weeks
  Ability of Gastrus to prevent and control gut microbiota alteration. Fecal samples for microbiological analysis will be collected before PPI treatment and at week 4, week 10 (end of PPI treatment) and week 14 (4 weeks after PPI discontinuation). The gas-chromatography mass spectrometry-solid-phase microextraction (GC-MS/SPME) analysis of fecal volatile compounds will be also performed.
Gastrointestinal Symptom Rating Scale (GSRS). | 14 weeks
  Participants will be asked to fill out the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire after inclusion but before taking the first dose of study product, every 2 weeks during treatment, and 2 weeks after stopping PPI. The GSRS is composed by 15 items combine into five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. Subjects rated the relevance and importance of each of the 15 GSRS items using the following scale:
  0 = Totally irrelevant
  1. = Relevant but not important
  2. = Moderately important
  3. = Very important Higher scores indicate greater severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Fernanda, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided
we will decide

REFERENCES:
- [Result] Kahrilas PJ, Shaheen NJ, Vaezi MF, Hiltz SW, Black E, Modlin IM, Johnson SP, Allen J, Brill JV; American Gastroenterological Association. American Gastroenterological Association Medical Position Statement on the management of gastroesophageal reflux disease. Gastroenterology. 2008 Oct;135(4):1383-1391, 1391.e1-5. doi: 10.1053/j.gastro.2008.08.045. No abstract available. PMID 18789939
- [Result] Wandall JH. Effects of omeprazole on neutrophil chemotaxis, super oxide production, degranulation, and translocation of cytochrome b-245. Gut. 1992 May;33(5):617-21. doi: 10.1136/gut.33.5.617. PMID 1319381
- [Result] DELLIPIANI AW, GIRDWOOD RH. BACTERIAL CHANGES IN THE SMALL INTESTINE IN MALABSORPTIVE STATES AND IN PERNICIOUS ANAEMIA. Clin Sci. 1964 Jun;26:359-74. No abstract available. PMID 14191265